CLINICAL TRIAL: NCT06524973
Title: Impacting Quality of Life and Pancreatic Cancer Survivorship Through a Telehealth Intervention
Brief Title: Telehealth Self-Management Coaching Sessions to Improve Quality of Life in Pancreatic Cancer Survivors and Their Family Care Givers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24172; NCI-2024-06078 (Other: P30)
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — Telemedicine; Counseling; Practice Guidelines as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (telehealth self-management coaching sessions) (Experimental): Patients and FCGs attend telehealth self-management coaching sessions over 40-60 minutes every other week for 6 sessions over 3 months.
  Interventions: Other: Telemedicine; Other: Counseling; Other: Questionnaire Administration; Other: Inrweview
- Arm B (standard of care) (Active Comparator): Patients and FCGs receive standard of care on study.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Telemedicine — Attend telehealth self-management coaching sessions
  Arms: Arm A (telehealth self-management coaching sessions)
Other: Counseling — Attend telehealth self-management coaching sessions
  Arms: Arm A (telehealth self-management coaching sessions)
Other: Best Practice — Receive standard of care
  Arms: Arm B (standard of care)
Other: Questionnaire Administration — Ancillary studies
Other: Inrweview — Ancillary studies
  Arms: Arm A (telehealth self-management coaching sessions)

SUMMARY:
This clinical trial evaluates the impact of telehealth self-management coaching sessions on quality of life in pancreatic cancer survivors and their family care givers (FCGs). Patients with pancreatic cancer experience many symptoms because of the disease and treatment, which can have a negative impact on quality of life. Patients and their families have unmet needs during treatment, including a lack of quality of life programs that offer support to patients. Supporting patients and families on managing the physical symptoms, emotional well-being, social well-being and spiritual well-being with telehealth self-management coaching sessions may help improve quality of life, manage symptoms from treatment, and support families in their role as caregivers during treatment.

ELIGIBILITY:
Inclusion Criteria:

* • PATIENT: Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines

    * PATIENT: Age: ≥ 18 years
    * PATIENT: Eastern Cooperative Oncology Group (ECOG) ≤ 2
    * PATIENT: Ability to read and understand English or Spanish for questionnaires
    * PATIENT: Subjects must have histologically or cytologically confirmed diagnosis of metastatic pancreatic adenocarcinoma who are within 8 weeks of initial diagnosis
    * FAMILY CARE GIVER: Documented informed consent of the participant and/or legally authorized representative
  * Assent, when appropriate, will be obtained per institutional guidelines

    * FAMILY CARE GIVER: Age: ≥ 18 years
    * FAMILY CARE GIVER: Ability to read and understand English or Spanish for questionnaires
    * FAMILY CARE GIVER: A family member or friend identified by the patient and defined as a person who knows the patient well and is involved in the patient's medical care

Exclusion Criteria:

* • An employee who is under the direct/ indirect supervision of the principal investigator (PI)/ a co-investigator/ the study manager

  * A direct study team member

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2027-05-03 (Estimated); Study Completion 2027-05-03 (Estimated)

PRIMARY OUTCOMES:
Patient reported quality of life (QOL) | At baseline and at 3 months post randomization
  Patient reported quality of life will be assessed by the Functional Assessment of Cancer Therapy- Hepatobiliary (FACT-Hep) quality of life score. The primary analysis will be a treatment group comparison of the QOL at 3 months via linear regression model, with adjustment for baseline FACT-Hep score and stratification factors. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures. The dependent variables will be transformed to approximate normality as appropriate.

SECONDARY OUTCOMES:
Enrollment rate | Up to 25 months
  Feasibility of the intervention will be defined as at least 60% of eligible participants enrolling. Descriptive statistics will be used to summarize the feasibility of the intervention. Reasons for non-participation will be recorded and used to make needed modifications for improvement in future studies.
Intervention completion rate | Up to 6 months
  Feasibility of the intervention will be defined as at least 60% of participants completing ≥ 80% of the intervention (4 of 6 sessions). Descriptive statistics will be used to summarize the feasibility of the intervention. Reasons for attrition will be recorded and used to make needed modifications for improvement in future studies.
Rate of participants completing any follow-up assessments | Up to 6 months
  Feasibility of the intervention will be defined as at least 60% of participants completing any follow-up assessments after randomization. Descriptive statistics will be used to summarize the feasibility of the intervention. Reasons for attrition will be recorded and used to make needed modifications for improvement in future studies.
Participant experience | Up to 6 months
  Participant experiences with the intervention will be explored through qualitative data (structured exit interviews) from participants randomized to the intervention group and analyzed using content analysis approach. Interviews will be transcribed and data analyzed. Transcripts will be imported for the development of analytic categories, data coding, and review of coded data. Codes will be sorted into themes based on links and relationship.
Patient reported symptom severity | At baseline and at 3 and 6 months post randomization
  Treatment group comparisons will be assessed via repeated measures linear regression models with adjustment for baseline value of the outcome including sex and age and stratification factors. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures. The dependent variables will be transformed to approximate normality as appropriate.
Patient reported psychological distress | At baseline and at 3 and 6 months post randomization
  Patient reported psychological distress will be measured using the National Comprehensive Cancer Network (NCCN) Distress Thermometer (DT). Treatment group comparisons will be assessed via repeated measures linear regression models with adjustment for baseline value of the outcome including sex and age and stratification factors. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures. The dependent variables will be transformed to approximate normality as appropriate.
Family care giver (FCG) psychological distress | At baseline and at 3 and 6 months post randomization
  FCG reported psychological distress will be measured using the NCCN DT. Treatment group comparisons will be assessed via repeated measures linear regression models with adjustment for baseline value of the outcome including sex and age and stratification factors. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures. The dependent variables will be transformed to approximate normality as appropriate.
FCG caregiving burden | At baseline and at 3 and 6 months post randomization
  FCG caregiving burden will be measured using the Montgomery Borgatta Caregiver Burden Scale. Treatment group comparisons will be assessed via repeated measures linear regression models with adjustment for baseline value of the outcome including sex and age and stratification factors. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures. The dependent variables will be transformed to approximate normality as appropriate.
FCG QOL | At baseline and at 3 and 6 months post randomization
  FCG QOL will be measured using City of Hope Quality of Life-Family questionnaire. Treatment group comparisons will be assessed via repeated measures linear regression models with adjustment for baseline value of the outcome including sex and age and stratification factors. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures. The dependent variables will be transformed to approximate normality as appropriate.
Overall survival | From initiation of intervention to death from any cause, up to 6 months

OTHER OUTCOMES:
Chemotherapy in last 14 days of life | At 3 and 6 months post randomization
Emergency room visits in the last days of life | At 3 and 6 months post randomization
Intensive care unit admissions in the last 30 days of life | At 3 and 6 months post randomization
Hospice care for less than 3 days before death | At 3 and 6 months post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chung, MD, Principal Investigator — City of Hope Medical Center
Locations (22):
- United States (22):
  - City of Hope at Arcadia, Arcadia, California
  - City of Hope Corona, Corona, California
  - City of Hope at Duarte, Duarte, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Glendale, Glendale, California
  - City of Hope at Glendora, Glendora, California
  - City of Hope Seacliff, Huntington Beach, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope at Irvine Sand Canyon, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope at Long Beach Worsham, Long Beach, California
  - City of Hope at Long Beach Elm, Long Beach, California
  - City of Hope Mission Hills, Mission Hills, California
  - City of Hope at Newport Beach Fashion Island, Newport Beach, California
  - City of Hope at Palmdale, Palmdale, California
  - City of Hope - Santa Clarita, Santa Clarita, California
  - City of Hope at Simi Valley, Simi Valley, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope at Thousand Oaks, Thousand Oaks, California
  - City of Hope South Bay, Torrance, California
  - City of Hope Upland, Upland, California
  - City of Hope West Covina, West Covina, California

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided